CLINICAL TRIAL: NCT06032819
Title: Artificial Intelligence for Differentiating Between Brain Hemorrhage and Contrast Extravasation After Mechanical Revascularization in Acute Ischemic Stroke
Brief Title: Differentiating Between Brain Hemorrhage and Contrast
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Hong Kong University of Science and Technology (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); The Seventh Affiliated Hospital of Sun Yat-sen University (Other); Peking University Shenzhen Hospital (Other); The Third Affiliated Hospital of Guangzhou Medical University (Other); The Third Affiliated Hospital of Southern Medical University (Other Government); Shenshan Medical Center, Memorial Hospital of Sun Yat-sen University (Unknown); Shantou Central Hospital (Other); Dongguan People's Hospital (Other Government); The First People's Hospital of Qinzhou (Unknown); Guangdong 999 Brain Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-865-01
Record Dates: First submitted 2023-09-04; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Ischemic Stroke
Keywords: Hemorrhage; Contrast Media Extravasation; Artificial Intelligence; Mechanical Revascularisation
MeSH Terms: conditions — Ischemic Stroke; Hemorrhage; Extravasation of Diagnostic and Therapeutic Materials

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hemorrhage: The result of the Intracranial hyper-density on CT images is determined by dual-energy CT or follow-up images: hyper-density can be seen on the virtual non-contrasted image of dual-energy CT, or high density persist longer than 48 hours.
- simple contrast extravasation: There is no Intracranial hyper-density on the virtual non-contrast images of dual-energy CT, or the follow-up CT show that the hyper-density is absorbed within 48 hours.

SUMMARY:
The goal of this observational study is to use artificial intelligence to differentiate cerebral hemorrhage from contrast agent extravasation after mechanical revascularization in ischemic stroke.

The main question it aims to answer is: Whether artificial intelligence can help differentiate brain hemorrhage from contrast agent extravasation.

Patients with intracranial high-density lesions on CT scans within 24h after mechanical revascularization will be included. Expected to enroll 500 patients. The type of high-density lesion is determined according to dual-energy CT images or follow-up images. Patients will be divided into training group, validation and testing groups by stratified random sampling (6:2:2). After the images and the image labels are obtained, deep learning artificial intelligence will be used to learn the image characteristics and establish a diagnostic model, and the model performance and generalization ability will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

(1) patients underwent non-enhanced head CT after mechanical vascularization; (2) initial post-operative non-enhanced head CT was performed within 24 h after mechanical vascularization; and (3) intracranial hyper-intensity, which was defined as an objectively higher density than the surrounding grey or white matter in the parenchyma or higher density than cerebrospinal fluid in ventricles and cisterns, could be seen on the initial non-enhanced head CT after mechanical vascularization.

Exclusion Criteria:

(1) the follow-up time of non-enhanced head CT after mechanical vascularization was less than 24 h; (2) artifacts (e.g. metal artifacts or motion artifacts) affected the hyper-intensity in CT images; and (3) patients underwent craniotomy after mechanical vascularization, which made it difficult to identify the area of hyper-intensity.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From December 2017 to June 2023, patients with acute ischemic stroke or intracranial arterial stenosis who underwent mechanical vascularization at 10 centers will be retrospectively enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Develop a deep learning model to differentiate brain hemorrhage from contrast agent extravasation, and evaluate the model performance and generalization ability | 2024-12
  The accuracy, sensitivity, specificity, precision, and recall of the model will be calculated, and confusion matrix will be display.

IPD SHARING:
Plan to Share IPD: Undecided